CLINICAL TRIAL: NCT01847690
Title: Effect of Cortisol on Physical Exertion in Patients With Primary Adrenal
Brief Title: Effect of Cortisol on Physical Exertion in Patients With Primary Adrenal Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/2216; 2012-005117-40 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-05-07 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Addison Disease
Keywords: Addison Disease
MeSH Terms: conditions — Addison Disease | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Treatment B is placebo (2 placebo tablets).
- Hydrocortisone (Active Comparator): Treatment A is 10 mg hydrocortisone (2 tablets Cortef, 5 mg each),Stress-dose will be taken per os one time 2 tablets 10 mg of Cortef 60 min before start of exercise. Cortef tablets 5 mg produced by Pharmacia and Upjohn . One day.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Cortef 5 mg tablets per os, 2x5 mg, one day, one time
  Other Names: Cortef
  Arms: Hydrocortisone

SUMMARY:
The conventional glucocorticoid replacement therapy in primary adrenal insufficiency- Addison's disease,renders the cortisol levels unphysiological, which may cause symptoms and long-term complications. Many patients take stress-doses that are extra doses of hydrocortisone or cortisone acetate before or during stressful physical or psychological events. However, the effect of such dosing has not been tested in scientific studies. In this double blind cross-over designed pilot trial we aim to test the effect of an extra dose of cortisol on physical activity and hormone levels.

DETAILED DESCRIPTION:
Addison's disease occurs when more than 90% of the adrenal cortex is destroyed. Cortisol levels in serum vary throughout the day. In addition to the daily need, cortisol increases in response to all forms of stress including intercurrent illness. The Addison patient must in such situations increase replacement doses 2 to 3-fold. While it is broad agreement on this procedure based on clinical experience and empirical data, it is controversial as to whether there is a need to increase the dose by less stressful events and tasks, such as average to vigorous physical activity and mental stress. In any event, many patients report that they benefit from stress doses not only in order to increase performance, but also to reduce post-exertion fatigue.

Using a combination of oxygen uptake measurements under controlled exercise and assay of hormones and metabolites, we aim to test whether extra doses of hydrocortisone can increase physical capacity and reduce post-exertion fatigue. Each patient perform two tests, one with and one without hydrocortisone in randomised order. The controls perform one test. The patients will be assigned a participation number and randomised to any of two treatment sequences (A-B or B-A) by pharmacy. All exercise tests will be performed 3-5 hours after intake of morning medication, after an overnight fast (water permitted). Patients will be instructed to avoid caffeinated food and drink, alcohol, strenuous exercise and starvation for at least 24h before each exercise session. Patients will be instructed to avoid smoking, brush teeth one hour before exercise testing.

One hour before each test, subjects drink one teaspoon of water per kilogram body weight to provide adequate hydration. Stress-dose or placebo will be taken 60 min before start. Also at this time, an indwelling line will be placed in the forearm of each subject that blood and saliva can be drawn before, directly after exercise, then 15 or 30 min after termination of exercise. Patients fill out the questionnaire about quality of life after each exercise.

Patient's daily glycemic profile will be followed up by continuous glucose monitoring systems for 24 hours before, during and for 24 hours after exercise. Patients will be educated in using the sensor and calibration with blood glucose self-measurements three to four times per day. Calibration of the sensor will be performed according to the protocol established. At the completion of the measuring period, the system will be returned, and the data will be downloaded to determine glucose patterns. This device will be applied to the abdomen of each subject, 24 h before each exercise session, calibrated as recommended (before operation and 2-3 additional times/day, 6 h apart over the 24 h of the study) and removed 24 h after the exercise session.

The patient's movements will be followed for 24 hour by Actigraph after each test. The test is repeated after 1 week with the opposite treatment option.

Ten adult patients (18-70 years) with verified Addison's disease will be invited to participate in the study. From a list of patients (consecutive out-patients or a patient registry) unselected patients should be invited to participate. Five age and sex matched healthy controls will be included to assess normal metabolic and endocrine responses to physical activity.

The investigator will keep a log of all patients that have been invited to participate in the study. If a screened patient does not fulfil the inclusion criteria, the reason will be documented on a screening log. Eligible patients who fulfil all of the inclusion criteria and none of the exclusion criteria will be randomised. Randomization will be performed by the hospital pharmacies at each study site. When a subject is randomized, he or she must always be assigned to the lowest available randomization number. The patients will be randomised in blocks of two to secure even patient number in each treatment sequence.

The patient will have to give written informed consent. The patients should not take grapefruit juice, liquorice and do not be on a special diet the last two weeks before or during the study period. Patients will be instructed to avoid caffeinated food and drink, alcohol, strenuous exercise and starvation for at least 24 h before each exercise session. Patients will be instructed to avoid smoking at least one hour before each exercise session.

Withdrawal criteria/Adverse Events. The patient is free to withdraw at any time. If a patient is having major difficulties managing the exercise the investigator will consider withdrawal. In the best interest of the patient, the investigator and the sponsor can decide to withdraw the patient from the study. If a patient develops conditions meeting the exclusion criteria, the patient will be withdrawn from the study. In case of serious adverse events the patient may be withdrawn from the study.

Any adverse event will be registered and reported to the Norwegian Medicines Agency. Any serious adverse events will be reported within 15 days, and in case of lethal or life threatening events immediately. The patients will report any problems or discomfort during or after examination in the patient log or diary, any need for extra doses during the study day after exercise with glucocorticoids will also be documented there. In addition, we ask them to contact the study group directly in case of problems between visits. The study documentation and research date will be stored 15 years after the termination of the study.

Statistical considerations This is a pilot study to evaluate the effect stress-dosing of cortisol on physical capacity. The results will be used for statistical calculations of effect size for a larger trial. The variation of the various efficacy parameters in this group of patients is not well known.

ELIGIBILITY:
Inclusion Criteria:

* patients with Addison's disease

Exclusion Criteria:

* Type 1 diabetes
* malignant disease
* pregnant women
* cardiac disease
* lung disease
* neuromuscular diseases
* pharmacological treatment with glucocorticoids or drugs that interfere with cortisol metabolism (anti-epileptics, rifampicin, St Johns wart, oral estrogens, antidepressives).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
O2 uptake | 2 days
  O2 uptake as V O2 90%.

SECONDARY OUTCOMES:
post- exercise hypoglycemic events | 4 days
  blood glucose below ≤ 3.1 mmol ⁄ L
glycemic variability | 6 days
  glycemic variability monitored by continuous glucose monitoring system
hormone response to exercise | 2 days
  * Plasma norepinephrine, epinephrine, salivary alfa amylase
  * Glucose, insulin, C-peptide, and lactate, glucagon
  * Growth hormone and insulin like growth factor
  * Free fatty acids
Blood pressure | 2 days
  vascular action
Subjective health status | 2 days
  Self administration by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Eystein Husebye, Professor, Study Director — Haukeland University Hospital; Katerina Simunkova, MUDr. PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland Universitetessykehus, Department of Medicine, Bergen, Norway, Norway

REFERENCES:
- [Background] Neary N, Nieman L. Adrenal insufficiency: etiology, diagnosis and treatment. Curr Opin Endocrinol Diabetes Obes. 2010 Jun;17(3):217-23. doi: 10.1097/MED.0b013e328338f608. PMID 20375886
- [Background] Weise M, Drinkard B, Mehlinger SL, Holzer SM, Eisenhofer G, Charmandari E, Chrousos GP, Merke DP. Stress dose of hydrocortisone is not beneficial in patients with classic congenital adrenal hyperplasia undergoing short-term, high-intensity exercise. J Clin Endocrinol Metab. 2004 Aug;89(8):3679-84. doi: 10.1210/jc.2003-032051. PMID 15292287
- [Background] Wurtman RJ, Axelrod J. Control of enzymatic synthesis of adrenaline in the adrenal medulla by adrenal cortical steroids. J Biol Chem. 1966 May 25;241(10):2301-5. No abstract available. PMID 4287854
- [Background] Ehrhart-Bornstein M, Bornstein SR. Cross-talk between adrenal medulla and adrenal cortex in stress. Ann N Y Acad Sci. 2008 Dec;1148:112-7. doi: 10.1196/annals.1410.053. PMID 19120098
- [Background] Bornstein SR, Breidert M, Ehrhart-Bornstein M, Kloos B, Scherbaum WA. Plasma catecholamines in patients with Addison's disease. Clin Endocrinol (Oxf). 1995 Feb;42(2):215-8. doi: 10.1111/j.1365-2265.1995.tb01866.x. PMID 7704967
- [Background] Green-Golan L, Yates C, Drinkard B, VanRyzin C, Eisenhofer G, Weise M, Merke DP. Patients with classic congenital adrenal hyperplasia have decreased epinephrine reserve and defective glycemic control during prolonged moderate-intensity exercise. J Clin Endocrinol Metab. 2007 Aug;92(8):3019-24. doi: 10.1210/jc.2007-0493. Epub 2007 May 29. PMID 17535996
- [Background] Weise M, Mehlinger SL, Drinkard B, Rawson E, Charmandari E, Hiroi M, Eisenhofer G, Yanovski JA, Chrousos GP, Merke DP. Patients with classic congenital adrenal hyperplasia have decreased epinephrine reserve and defective glucose elevation in response to high-intensity exercise. J Clin Endocrinol Metab. 2004 Feb;89(2):591-7. doi: 10.1210/jc.2003-030634. PMID 14764767
- [Background] Merke DP, Chrousos GP, Eisenhofer G, Weise M, Keil MF, Rogol AD, Van Wyk JJ, Bornstein SR. Adrenomedullary dysplasia and hypofunction in patients with classic 21-hydroxylase deficiency. N Engl J Med. 2000 Nov 9;343(19):1362-8. doi: 10.1056/NEJM200011093431903. PMID 11070100
- See also: endocrine society — http://www.ese-hormones.org